CLINICAL TRIAL: NCT02967185
Title: Intraindividual Variability in Sleep and Cognitive Performance in Older Adults
Acronym: REST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: University of Florida (Other)
Responsible Party: Principal Investigator, Christina McCrae, Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 221286
Record Dates: First submitted 2016-11-08; First posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Insomnia Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief Behavioral Therapy for Insomnia (Experimental): Treatment will consist of 4 weekly, 1 hour sessions and will be conducted by a trained graduate assistant on an individual basis.
  Interventions: Behavioral: Brief Behavioral Therapy for Insomnia
- Waitlist Control (No Intervention): Participants in this group will receive no intervention, but will complete the same set of assessments as those in the Experimental Group. They will be given the option of receiving the behavioral treatment program at no charge.

INTERVENTIONS:
Behavioral: Brief Behavioral Therapy for Insomnia — Treatment will consist of 4 weekly, 1 hour sessions and will be conducted by a trained graduate assistant on an individual basis. Treatment components will include education about aging and sleep. It will also include instruction in techniques designed to: (a) promote good sleep habits, (b) restrict the use of the bed and bedroom to sleep and sleep-conducive activities, (c) modify bed and wake times to better match the participants sleep needs, and (d) promote relaxation. Daily home practice of these techniques will be encouraged. Participants will maintain logs of their home practice sessions and will continue to record their daily sleep habits throughout treatment.
  Arms: Brief Behavioral Therapy for Insomnia

SUMMARY:
The proposed study will examine changes in older insomniacs' cognitive functioning following behavioral treatment for insomnia using a combination of two methods. A traditional repeated measures design will be used to look at group level differences based on performance on a neuropsychological battery administered prior to, immediately after, and 3 months after completing a 4 week behavioral treatment program for insomnia. This data will be analyzed using standard repeated measures analytic techniques. A time-series design will also be used to look at within-subject differences based on a brief cognitive battery that will be self-administered on a daily basis. Data from this daily battery will be examined using intraindividual variability modeling.

ELIGIBILITY:
Inclusion Criteria:

* Age >65 years
* Community dwelling
* Available for duration of study
* Insomnia according to American Sleep Disorders Association (1990) criteria: (a) >30 minutes of unwanted awake time, 3 nights per week for at least 6 months and (b) Daytime dysfunction (reported mood, cognitive, social, or occupational impairment)

Exclusion Criteria:

* Age less than 65
* history of primary sleep disorder (e.g., sleep apnea, narcolepsy)
* history of stroke
* major medical illness known to contribute to sleep problems in last 12 months
* cognitive impairment that interferes with ability to understand treatment (score <23 on Mini-Mental State Examination)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2005-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Change in diary-assessed total sleep and wake time during sleep from baseline to follow-up | from baseline to follow-up, approximately 1 year
  Participants will complete a daily sleep dairies throughout the study period. They will report their bedtime, waketime, sleep onset latency, and wake time after sleep onset. Total sleep time and total wake time will be calculated from the diaries.

SECONDARY OUTCOMES:
Change in actigraphy-assessed sleep variability from baseline to follow-up | from baseline to follow-up, approximately 1 year
  Participants wore an Actiwatch-L (ACTL) (Mini Mitter Co., Inc.) on their non-dominant wrists continuously throughout the study. The sensor of the ACTL is sampled 32 times per second and records peak values for each second. These peak values are then summed into 30-second "activity" counts. These activity counts are downloaded to a personal computer and analyzed using Actiware-Sleep v. 3.3, which uses a validated algorithm to identify periods of as sleep or wake. Total sleep time and total wake time will be computed.
Change in performance on the Mini-Mental Status Exam | from baseline to follow-up, approximately 1 year
  Mini-Mental Status Exam (MMSE) (Folstein, Folstein, & McHugh, 1975)
Change in performance on Wechsler Adult Intelligence Scale-3, Vocabulary & Digit Symbol | from baseline to follow-up, approximately 1 year
  Wechsler Adult Intelligence Scale-3, Vocabulary & Digit Symbol (subtests) [WAIS-3]
Change in performance on the Trails A & B (Reitan, 1958) | from baseline to follow-up, approximately 1 year
  Trails A & B (Reitan, 1958) was administered
Change in performance on the Controlled Oral Word Association | from baseline to follow-up, approximately 1 year
  Controlled Oral Word Association (COWA) (Benton & Hamsher, 1983)
Change in performance on the Boston Naming Test (BNT) | from baseline to follow-up, approximately 1 year
  Boston Naming Test (BNT)
Change in performance on the California Verbal Learning Test (CVLT, CVLT-II) | from baseline to follow-up, approximately 1 year
  California Verbal Learning Test (CVLT, CVLT-II) (Delis, Kramer, Kaplan, & Ober, 1987)
Change in performance on the Rey-Osterreith Complex Figure Test (Rey-O) (Hubley & Tremblay, 2002) | from baseline to follow-up, approximately 1 year
Change in performance on the Wechsler Memory Scale-3, Logical Memory & Visual Reproduction subtests (WMS-3) Tremblay, 2002) | from baseline to follow-up, approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christina McCrae, PhD, Principal Investigator — University of Missouri-Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McCrae CS, McGovern R, Lukefahr R, Stripling AM. Research Evaluating Brief Behavioral Sleep Treatments for Rural Elderly (RESTORE): a preliminary examination of effectiveness. Am J Geriatr Psychiatry. 2007 Nov;15(11):979-82. doi: 10.1097/JGP.0b013e31813547e6. PMID 17974868
- [Derived] McCrae CS, Curtis AF, Williams JM, Dautovich ND, McNamara JPH, Stripling A, Dzierzewski JM, Berry RB, McCoy KM, Marsiske M. Effects of Brief Behavioral Treatment for Insomnia on Daily Associations between Self-Reported Sleep and Objective Cognitive Performance in Older Adults. Behav Sleep Med. 2020 Sep-Oct;18(5):577-588. doi: 10.1080/15402002.2019.1632201. Epub 2019 Jun 15. PMID 31203649
- [Derived] Curtis AF, Williams JM, McCoy KJM, McCrae CS. Chronic Pain, Sleep, and Cognition in Older Adults With Insomnia: A Daily Multilevel Analysis. J Clin Sleep Med. 2018 Oct 15;14(10):1765-1772. doi: 10.5664/jcsm.7392. PMID 30353817
- [Derived] McCrae CS, Curtis AF, Williams JM, Dautovich ND, McNamara JPH, Stripling A, Dzierzewski JM, Chan WS, Berry RB, McCoy KJM, Marsiske M. Efficacy of brief behavioral treatment for insomnia in older adults: examination of sleep, mood, and cognitive outcomes. Sleep Med. 2018 Nov;51:153-166. doi: 10.1016/j.sleep.2018.05.018. Epub 2018 Jun 2. PMID 30195661
- [Derived] Chan WS, Williams J, Dautovich ND, McNamara JPH, Stripling A, Dzierzewski JM, Berry RB, McCoy KJM, McCrae CS. Night-to-Night Sleep Variability in Older Adults With Chronic Insomnia: Mediators and Moderators in a Randomized Controlled Trial of Brief Behavioral Therapy (BBT-I). J Clin Sleep Med. 2017 Nov 15;13(11):1243-1254. doi: 10.5664/jcsm.6790. PMID 28992829